CLINICAL TRIAL: NCT04219293
Title: A Single-center, Randomized, Split Face Study of the Effects of Micro Needling With Platelet Rich Plasma Compared to Microneedling Without Platelet Rich Plasma
Brief Title: Split Face Study of the Effects of Micro Needling With and Without Platelet Rich Plasma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-19
Sponsor: Dallas Plastic Surgery Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: PRP01
Record Dates: First submitted 2019-12-09; First posted 2020-01-07 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Aging

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Microneedling with NO PRP (Other): Patient will receive Standard of Care micro needling on randomized side of the face.
  Interventions: Device: Microneedling w/ and w/o PRP
- Microneedling WITH PRP (Active Comparator): Patient will receive Standard of care microneedling with PRP on randomized side of the face.
  Interventions: Device: Microneedling w/ and w/o PRP

INTERVENTIONS:
Device: Microneedling w/ and w/o PRP — i. Split face comparison. Vertical line drawn midline nose extending upwards to hairline and downwards to jawline separating face into two equal treatment areas. The patients determined side of face will be treated with SkinPen Microneedling and PRP the other (nondetermined from randomization) will be treated with SkinPen Microneedling and glide. The patient side of face that will not use PRP will be treated first. The following settings will be used as treatment protocol. Topical anesthetic Benzocaine 20%, Lidocaine 10%, and Tetracaine 10% will be applied covering entire treatment area. The anesthetic will remain on skin for 30 minutes.

SUMMARY:
This pilot study will expand knowledge and application of 2 X concentration of Platelet Rich Plasma (PRP) in conjunction with microneedling using the SkinPen device.

DETAILED DESCRIPTION:
There have been numerous studies demonstrating benefits of microneedling. However, to date there is no published research expanding on the benefits of using platelet rich plasma in conjunction with microneedling for facial aesthetics. This pilot study will expand knowledge and application of 2 X concentration of Platelet Rich Plasma (PRP) in conjunction with microneedling using the SkinPen device. The pilot aims to objectively measure skin quality using the Visia systemTM and provide objective data to compare Microneedling with the use of (PRP) versus microneedling without the use of PRP. The pilot also aims to subjectively measure skin improvement using the Face QTM and the Global Aesthetic Improvement ScaleTM.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females ages 30-60 years old.
* No previous minimally invasive or invasive skin resurfacing within the prior 12 months (i.e. fractionated laser, ablated laser, chemical peels, microneedling, etc…
* VisiaTM Scan showing aging including skin texture, wrinkles, brown spots, and pores.
* Patient willing to sign informed consent.

Exclusion Criteria:

* Keloid scars;
* History of eczema in treatment area; psoriasis and any other chronic skin conditions the Investigator determines disqualifies the patient for participation in treatment area;
* History of actinic (solar) keratosis in treatment area;
* History of hemophilia;
* History of diabetes;
* The presence of raised moles, warts on the targeted area.
* Absolute contraindications include; scleroderma, collagen vascular diseases or cardiac abnormalities; blood clotting problems; active bacterial or fungal infection; facial melanosis; malignant tumors, immunosuppression; use of blood thinners or prednisone; pregnant or nursing women; corticosteroids within two weeks of the procedure, chronic liver disease, porphyria or other skin diseases.
* Patient not willing to sign informed consent.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Overall Skin improvement assessed by a Visia Scan. | 6 months
  The VISIA® facial scan uses 3-D imaging to accurately identify and quantify all aesthetic skin concerns, even before there are visible signs of damage or aging. Using a state-of-the-art, multi-point positioning system the visia scanner captures multiple angles of your skin.
Overall Patient satisfaction of skin improvement assessed by the Global Aesthetic Improvement Scale. | 6 months
  The Global Aesthetic Improvement Scale (GAIS) is a 5-point scale rating global aesthetic improvement in appearance, compared to pretreatment, as judged by the investigator.
Overall Patient satisfaction of skin improvement assessed by the Face-Q Aesthetic Satisfaction with Outcome. | 6 months
  The FACE-Q© is a patient-reported outcome (PRO) measure that can be used to measure outcomes of. aesthetic facial procedures and products from the patient's perspective.
Overall Patient satisfaction of skin improvement assessed by the Face-Q Aesthetic Satisfaction with Skin. | 6 months
  The FACE-Q© is a patient-reported outcome (PRO) measure that can be used to measure outcomes of. aesthetic facial procedures and products from the patient's perspective.

CONTACTS AND LOCATIONS:
Locations (1):
- Dallas Plastic Surgery Institute, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No